CLINICAL TRIAL: NCT00584571
Title: Randomized Controlled Trial of Treating Rectal Hypersensitivity - Comparing Escitalopram With Sensory Adaptation Training
Brief Title: SAT vs Escitalopram for Rectal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2R01 KD57100-05A2; 2R01DK057100-06A2 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Rectal Hypersensitivity; Irritable Bowel Syndrome-Constipation
MeSH Terms: interventions — Escitalopram; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensory Adaptation training (Active Comparator): a large compliant balloon is placed in the rectum attached to a barostat. The balloon is distended in 1 mm increments until patient reports moderate discomfort and then increased in 1 mm increments until maximum tolerable pressure. Gradually over 6 training sessions, administered biweekly, the maximum tolerable pressure is increased over 3 months, if treatment is successful.
  Interventions: Procedure: Sensory Adaptation Training
- Escitalopram Therapy (Experimental): Patients randomized to this arm will receive daily 10 mg escitalopram for 3 months. If the medication is effective their bowel symptoms and pain thersholds will improve.
  Interventions: Drug: Escitalopram Therapy

INTERVENTIONS:
Procedure: Sensory Adaptation Training — This study will last for approximately 3 months and will include 4-6 clinic visits with each visit lasting 2 hours every week or every 2 weeks. At the beginning of each visit we will ask you about your health status and level of satisfaction of your bowel habits. We will then place the pencil-thick probe and balloon inside your rectum and attach it to the barostat device and a computer. We will increase and decrease the volumes of the balloon until the most pressure you can tolerate or a certain level of pressure as measured by the machine is reached, whichever occurs first. You will continue to keep stool diaries and pain diaries for 7 days before and after each visit.
  Other Names: Barostat procedure
  Arms: Sensory Adaptation training
Drug: Escitalopram Therapy — Escitalopram; 10 mg every day, orally.
  Other Names: Lexapro (Escitalopram) therapy
  Arms: Escitalopram Therapy

SUMMARY:
Constipation is a common digestive disorder. After excluding dietary factors, drugs and other secondary causes, at least three broad pathophysiologic subtypes are recognized- dyssynergic defecation, constipation-predominant irritable bowel syndrome (IBS-C) and slow transit constipation (STC), all predominantly affect women and elderly. Many patients also demonstrate abnormal rectal perception with both rectal hyposensitivity and hypersensitivity being common. Recent surveys show that most constipated patients are dissatisfied with current therapy. Also, constipated patients showed significant psychological dysfunction and impaired quality of life. OBJECTIVE: To investigate a novel biofeedback technique of improving rectal hypersensitivity.

METHODS: A large compliant balloon attached to a barostat was placed in the rectum in 8 patients with rectal hypersensitivity (urgency/pain threshold <30 mm Hg). Sensory deconditioning was performed by incremental balloon distensions (1-2 mmHg) until normal thresholds were reached.

DETAILED DESCRIPTION:
To investigate a novel biofeedback technique of improving rectal hypersensitivity using rectal barostat and to compare this with clinical standard of care comprising of low dose antidepressant therapy with escitalopram. Patients will be randomized to sensory adaptation training or escitalopram in a 1:1 ratio

ELIGIBILITY:
Inclusion Criteria:

All patients must fulfill the diagnostic criteria for IBS-C (Rome III) as defined below and have rectal hypersensitivity (see below).

* Patients must report recurrent abdominal pain or discomfort for at least 3 days per month in the last 3 months with two or more of the following symptoms:

  * Improvement with defecation; and/or
  * Onset associated with a change in frequency of stool; and/or
  * Onset associated with a change in form (appearance) of stool
* No structural diseases
* On a diary:

  * Pain/discomfort for at least 2 days/week;
  * No loose or watery stool <25% of bowel movements.

Exclusion Criteria:

* Patients with mixed-IBS.
* Patients currently on SSRI or MAO inhibitors. Patients on stable doses of other antidepressants will be included provided the dose is unchanged during study.
* Patients taking drugs that are constipating, (e.g.; calcium channel antagonists will either be excluded or drug discontinued)
* Patients with co-morbid illnesses; severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy.
* Neurologic diseases e.g.; head injury, epilepsy, multiple sclerosis, strokes, spinal cord injuries.
* Impaired cognizance (mini mental score of < 15) and/or legally blind.
* Pregnant or likely to conceive during the course of the study. Women with potential for pregnancy must be willing to use contraceptive measures during the study. Urinary pregnancy tests will be performed on such women prior to any radiologic procedures.
* Hirschsprung's disease.
* Alternating constipation and diarrhea (22).
* Ulcerative/Crohns colitis.
* Previous pelvic surgery, rectocele/bladder repair, radical hysterectomy, anal surgery.
* Rectal prolapse or anal fissure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rectal Sensory Thresholds | Trial entry and at the end of 3 months
  The primary physiologic outcome measure is increase in rectal sensory thresholds after treatment. A rectal hypersensitivity responder is defined as an individual who show at least 20% increase in two or more sensory thresholds (first, desire and urge defecate/pain) after treatment when compared to baseline, and will be compared between the SAT and escitalopram groups. An overall responder is defined as both a hypersensitivity responder and abdominal pain responder.
Abdominal Pain | Trial entry and at the end of 3 months
  The symptomatic outcome measure is decrease in pain score as assessed by daily pain logs where pain is scored on a scale of 0 to 4, after treatment when compared to the baseline period. A pain responder is defined as a subject with 30% decrease in pain compared to baseline.

SECONDARY OUTCOMES:
Global Bowel Satisfaction Score (GSA) | Trial entry and at the end of 3 months
  The global bowel satisfaction will be analysed using a visual analog scale 0-10 cm (0 - very dissatisfied, 10 - completely satisfied).
Bowel symptoms | Trial entry and at the end of 3 months
  We will assess the number of complete spontaneous bowel movements, mean straining scores, mean stool consistency (Bristol Stool Scale) (numerical mean scores for individual questions) between the two groups.
Rectal compliance | Trial entry and at the end of 3 months
  We will assess the changes in intrarectal pressures and intrarectal volumes during Barostat rectal balloon distention between the two groups.
IBS quality of life | Trial entry and at the end of 3 months
  The IBS quality of life will be assessed using the 8 domains of IBS-QOL and compared between the two groups.
Psychological profiles | Trial entry and at the end of 3 months
  The psychological profiles will be assessed using the SCL-90R questionnaire and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Satish SC Rao, MD, PhD, Principal Investigator — Augusta University
Locations (2):
- United States (2):
  - Augusta University, Augusta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa

REFERENCES:
- [Derived] Rao SSC, Coss-Adame E, Yan Y, Erdogan A, Valestin J, Ayyala DN. Sensory Adaptation Training or Escitalopram for IBS With Constipation and Rectal Hypersensitivity: A Randomized Controlled Trial. Clin Transl Gastroenterol. 2021 Jul 13;12(7):e00381. doi: 10.14309/ctg.0000000000000381. PMID 34254966